CLINICAL TRIAL: NCT03150251
Title: Glycemic and Insulinemic Response to Oats Soaked Overnight in Milk Compared to Cream of Rice in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1610
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Glycemic, Insulinemic, Subjective Appetite Responses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Overnight Oats (Experimental): 40 g of overnight oats
  Interventions: Other: Cereal - oats
- Soaked Cream of Rice (Placebo Comparator): 28.8 cream of rice
  Interventions: Other: Cereal - cream of rice
- Cooked Cream of Rice (Placebo Comparator): 28.8 cooked cream of rice
  Interventions: Other: Cereal - cream of rice

INTERVENTIONS:
Other: Cereal - oats — Consumption of one cereal in the beginning of each visit
  Other Names: Oats
  Arms: Overnight Oats
Other: Cereal - cream of rice — Consumption of one cereal in the beginning of each visit
  Other Names: Cream of Rice
  Arms: Cooked Cream of Rice; Soaked Cream of Rice

SUMMARY:
One objective of this study is to examine the blood glucose and serum insulin responses over 2hr elicited by oats soaked overnight in milk compared to Cream of Rice soaked overnight in milk and compared to Cream of Rice cooked in water. In addition a second objective of the study is to measure subjective ratings of hunger and fullness under the same conditions.

ELIGIBILITY:
Inclusion Criteria:

Male or non-pregnant females, 18-75 years of age, inclusive

* Body mass index (BMI) between 20.00 and 34.99 kg/m² inclusive at screening (visit 1).
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
* Normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Wolever, the president of GI Testing, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at screening.
* Change in body weight of >3.5kg within 4 weeks of the screening visit.
* Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
* Exposure to any non-registered drug product within 30 d prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Incremental area under the blood glucose curve | 0-2 hours

SECONDARY OUTCOMES:
incremental areas under the curve of blood glucose from 2-3h | 2-3 hours
incremental areas under the curve of blood glucose from 0-3h | 0-3 hours
incremental areas under the curve of insulin serum 0-2 hours | 0-2 hours
incremental areas under the curve of insulin serum 2-3 hours | 2-3 hours
incremental areas under the curve of insulin serum 0-3 hours | 0-3 hours
peak concentrations and peak rises of glucose and insulin | 0-3 hours
blood glucose and insulin concentrations and increments at each time point over a 3hr period | 0-3 hours
netAUC of the curves for fullness, hunger, desire to eat, prospective consumption and average appetite over 0-2hr and 0-3hr | 0-2 hour and 0-3 hours
self reports of fullness, hunger, desire to eat, prospective consumption and average appetite at each point in time via questionnaires | 3 hours post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD, Principal Investigator — GI Laboratories
Locations (1):
- Glycemic Index Laboratories, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No